CLINICAL TRIAL: NCT06936839
Title: Optimal ECMO Flow in the Critical Phase of Cardiogenic Shock to Optimize Peripheral Organ Perfusion and Myocardial Stress
Acronym: ECMO-FLOW
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0215
Record Dates: First submitted 2025-03-26; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Cardiogenic Shock
Keywords: ECMO; optimal flow; cardiogenic shock; echocardiography; organ perfusion; myocardial recovery; human; adult; left ventricular overload
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study cohort: Adult patients at the early phase of a cardiogenic shock treated with veno-arterial ECMO (<48h)
  Interventions: Other: Obversation

INTERVENTIONS:
Other: Obversation — Observing the optimal flow rate to reduce left ventricular stress and enhance peripheral organ perfusion during ramp tests (conducted at QECMO levels of 100%, 75%, 50%, and 25%, provided that SVO₂ remains >55% and NIRS rSO₂ remains >50%)

SUMMARY:
Veno-arterial ECMO (VA ECMO) is considered the ultimate lifesaving technique in refractory cardiogenic shock (CS). However, VA ECMO is associated with potentially serious adverse effects and complications. Many authors have demonstrated that VA ECMO increases left ventricular (LV) afterload, leading to increased LV stress, left ventricular end-diastolic pressure (LVEDP), and left atrial pressure (LAP). This pressure increase frequently results in pulmonary oedema and higher myocardial oxygen consumption. These complications are critical to patient survival and myocardial recovery and can lead to prolonged hospital stays and increased healthcare costs.

In the absence of clinical studies and strong recommendations, the optimized management of VA ECMO in clinical practice involves finding an ECMO flow that balances adequate organ perfusion with preserved ventricular ejection, while minimizing LV stress. Since the optimal flow changes with myocardial recovery, ramp tests are regularly performed to adjust ECMO flow.

To date, the optimized management of VA ECMO has been guided empirically. The aim of this study is to describe the consequences of variations in VA ECMO flow during the critical phase of cardiogenic shock on peripheral organ perfusion and LV stress. By analyzing the relationships between VA ECMO flow rate, peripheral perfusion, and myocardial stress, investigators aim to optimize flow settings-particularly by minimizing the potential complications of VA ECMO.

During the daily ramp tests, investigators plan to collect hemodynamic data (cardiac output, SvO₂, pulse pressure, EtCO₂, vasopressor and inotrope dosing), echocardiographic measurements, and organ perfusion indicators (NIRSS, CO₂ gap, respiratory quotient, lactate levels). Data will be collected on Day 1 (ECMO initiation), Day 2 (24 hours after ECMO initiation), and Day 3 (48 hours after ECMO initiation).

ELIGIBILITY:
Inclusion Criteria:

* cardiogenic shock
* treated with VA ECMO for less than 48hours

Exclusion Criteria:

* ECMO initiated for refractory cardiac arrest
* Cardiac arres prior to the cardiogenic shock with Low-Flow > 30 min
* Noradrenaline dose > 1μg/kg/min, vasopressin dose > 2IU/h, dobutamine dose > 15μg/kg/min, adrenaline dose > 1μg/kg/min, or unstabilized vasopressors or inotropes
* Post-cardiotomy cardiogenic shock
* Septic shock
* Left ventricular unloading by Impella (CP/5) or atrioseptostomy
* Atrial septal defect
* Ventricular septal defect
* Pregnant or breast-feeding women
* Patients protected by law (under guardianship or curatorship),
* Patient participating in another research study with an exclusion period still in progress
* Opposition to participation after having been informed
* Patient not affiliated to any health care system
* Patient unable to express non-opposition without available trusted person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cardiogenic shock treated with VA ECMO for less than 48 hours without any of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
optimal flow | Day 1 (ECMO initiation), Day 2 (24 hours after ECMO initiation), and Day 3 (48 hours after ECMO initiation).
  ECMO flow indexed to body surface area, defined as the flow with minimum PCWP (pulmonary capillary wedge pressure) and SvO2>55% at different times after ECMO start (Day 1, day 2 and day 3).

SECONDARY OUTCOMES:
optimal flow according to echocardiography | Day 1 (ECMO initiation), Day 2 (24 hours after ECMO initiation), and Day 3 (48 hours after ECMO initiation).
  ECMO flow indexed to body surface area, defined as the flow with minimum LVEDD (Left Ventricular End-Diastolic Diameter) and SvO2>55% at different times after ECMO start (Day 1, day 2 and day 3).
optimal flow according to the patient's native cardiac output | Day 1 (ECMO initiation), Day 2 (24 hours after ECMO initiation), and Day 3 (48 hours after ECMO initiation).
  ECMO flow indexed to body surface area, defined as the flow with optimized native cardiac output (measured or estimated by EtCO2 and arterial pulse pressure) at different times after ECMO start (Day 1, day 2 and day 3).
optimal flow in subgroup 1 (low pulse pressure) | Day 1 (ECMO initiation), Day 2 (24 hours after ECMO initiation), and Day 3 (48 hours after ECMO initiation).
  Optimal flow as defined by the primary outcome in patients with low arterial pulse pressure (<15mmHg) at different times after ECMO start (Day 1, day 2 and day 3).
optimal flow in subgroup 2 (normal pulse pressure) | Day 1 (ECMO initiation), Day 2 (24 hours after ECMO initiation), and Day 3 (48 hours after ECMO initiation).
  Optimal flow as defined by the primary outcome in patients with normal arterial pulse pressure (>15mmHg) at different times after ECMO start (Day 1, day 2 and day 3).
Correlation between flow and other perfusion indicators | Day 1 (ECMO initiation), Day 2 (24 hours after ECMO initiation), and Day 3 (48 hours after ECMO initiation).
  test the correlation between flow rate and tissue perfusion indicators (SvO2, NIRSS, Respiratory quotient, CO2 gap).

CONTACTS AND LOCATIONS:
Overall Officials: Aurore Ughetto, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostadal P, Mlcek M, Kruger A, Hala P, Lacko S, Mates M, Vondrakova D, Svoboda T, Hrachovina M, Janotka M, Psotova H, Strunina S, Kittnar O, Neuzil P. Increasing venoarterial extracorporeal membrane oxygenation flow negatively affects left ventricular performance in a porcine model of cardiogenic shock. J Transl Med. 2015 Aug 15;13:266. doi: 10.1186/s12967-015-0634-6. PMID 26275717
- [Background] Burkhoff D, Sayer G, Doshi D, Uriel N. Hemodynamics of Mechanical Circulatory Support. J Am Coll Cardiol. 2015 Dec 15;66(23):2663-2674. doi: 10.1016/j.jacc.2015.10.017. PMID 26670067
- [Background] Fuhrman BP, Hernan LJ, Rotta AT, Heard CM, Rosenkranz ER. Pathophysiology of cardiac extracorporeal membrane oxygenation. Artif Organs. 1999 Nov;23(11):966-9. doi: 10.1046/j.1525-1594.1999.06484.x. PMID 10564298
- [Background] Burkhoff D, Sagawa K. Ventricular efficiency predicted by an analytical model. Am J Physiol. 1986 Jun;250(6 Pt 2):R1021-7. doi: 10.1152/ajpregu.1986.250.6.R1021. PMID 3717375
- [Background] Mallat J, Pepy F, Lemyze M, Gasan G, Vangrunderbeeck N, Tronchon L, Vallet B, Thevenin D. Central venous-to-arterial carbon dioxide partial pressure difference in early resuscitation from septic shock: a prospective observational study. Eur J Anaesthesiol. 2014 Jul;31(7):371-80. doi: 10.1097/EJA.0000000000000064. PMID 24625464
- [Background] Mesquida J, Saludes P, Gruartmoner G, Espinal C, Torrents E, Baigorri F, Artigas A. Central venous-to-arterial carbon dioxide difference combined with arterial-to-venous oxygen content difference is associated with lactate evolution in the hemodynamic resuscitation process in early septic shock. Crit Care. 2015 Mar 28;19(1):126. doi: 10.1186/s13054-015-0858-0. PMID 25888382
- [Background] Routsi C, Vincent JL, Bakker J, De Backer D, Lejeune P, d'Hollander A, Le Clerc JL, Kahn RJ. Relation between oxygen consumption and oxygen delivery in patients after cardiac surgery. Anesth Analg. 1993 Dec;77(6):1104-10. doi: 10.1213/00000539-199312000-00004. PMID 8250298
- [Background] Vallet B, Teboul JL, Cain S, Curtis S. Venoarterial CO(2) difference during regional ischemic or hypoxic hypoxia. J Appl Physiol (1985). 2000 Oct;89(4):1317-21. doi: 10.1152/jappl.2000.89.4.1317. PMID 11007564
- [Background] Bakker J, Vincent JL, Gris P, Leon M, Coffernils M, Kahn RJ. Veno-arterial carbon dioxide gradient in human septic shock. Chest. 1992 Feb;101(2):509-15. doi: 10.1378/chest.101.2.509. PMID 1735281
- [Background] Mecher CE, Rackow EC, Astiz ME, Weil MH. Venous hypercarbia associated with severe sepsis and systemic hypoperfusion. Crit Care Med. 1990 Jun;18(6):585-9. doi: 10.1097/00003246-199006000-00001. PMID 2111753
- [Background] Groeneveld AB. Interpreting the venous-arterial PCO2 difference. Crit Care Med. 1998 Jun;26(6):979-80. doi: 10.1097/00003246-199806000-00002. No abstract available. PMID 9635634
- [Background] Faden H. Prophylactic antibiotics in pediatrics cardiovascular surgery: current practices. Ann Thorac Surg. 1981 Mar;31(3):211-3. doi: 10.1016/s0003-4975(10)60928-9. PMID 7212816
- [Background] Moller JE, Sionis A, Aissaoui N, Ariza A, Belohlavek J, De Backer D, Farber G, Gollmann-Tepekoylu C, Mebazaa A, Price S, Swol J, Thiele H, Hassager C. Step by step daily management of short-term mechanical circulatory support for cardiogenic shock in adults in the intensive cardiac care unit: a clinical consensus statement of the Association for Acute CardioVascular Care of the European Society of Cardiology SC, the European Society of Intensive Care Medicine, the European branch of the Extracorporeal Life Support Organization, and the European Association for Cardio-Thoracic Surgery. Eur Heart J Acute Cardiovasc Care. 2023 Jul 7;12(7):475-485. doi: 10.1093/ehjacc/zuad064. PMID 37315190
- [Background] Chiolero RL, Revelly JP, Leverve X, Gersbach P, Cayeux MC, Berger MM, Tappy L. Effects of cardiogenic shock on lactate and glucose metabolism after heart surgery. Crit Care Med. 2000 Dec;28(12):3784-91. doi: 10.1097/00003246-200012000-00002. PMID 11153615
- [Background] Khosravani H, Shahpori R, Stelfox HT, Kirkpatrick AW, Laupland KB. Occurrence and adverse effect on outcome of hyperlactatemia in the critically ill. Crit Care. 2009;13(3):R90. doi: 10.1186/cc7918. Epub 2009 Jun 12. PMID 19523194
- [Background] Valenza F, Aletti G, Fossali T, Chevallard G, Sacconi F, Irace M, Gattinoni L. Lactate as a marker of energy failure in critically ill patients: hypothesis. Crit Care. 2005;9(6):588-93. doi: 10.1186/cc3818. Epub 2005 Sep 28. PMID 16356243
- [Background] Laine GA, Hu BY, Wang S, Thomas Solis R, Reul GJ Jr. Isolated high lactate or low central venous oxygen saturation after cardiac surgery and association with outcome. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1271-6. doi: 10.1053/j.jvca.2013.02.031. Epub 2013 Sep 5. PMID 24011873
- [Background] Abrams D, Combes A, Brodie D. What's new in extracorporeal membrane oxygenation for cardiac failure and cardiac arrest in adults? Intensive Care Med. 2014 Apr;40(4):609-12. doi: 10.1007/s00134-014-3212-0. Epub 2014 Jan 29. No abstract available. PMID 24474528